CLINICAL TRIAL: NCT06532383
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBOCONTROLLED, SINGLE-DOSE ESCALATION STUDY TO EVALUATE THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF-07940369 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-07940369 Are Tolerated and Act in the Body in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C5381001; 2024-513467-47-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded (investigator- and participant-blinded), sponsor-open, placebo-controlled, 4-period, crossover, interleaving, first in human single ascending oral dose
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be assigned to receive study intervention according to the assigned treatment group from the randomization scheme. Investigators will remain blinded to each participant's assigned study intervention throughout the course of the study. In order to maintain this blind, an otherwise uninvolved third party will be responsible for the preparation and dispensing of all study intervention and will endeavor to ensure that there are no differences in time taken to dispense or visual presentation, following randomization or dispensing. This third party will instruct the participant to avoid discussing the taste, dosing frequency, or packaging of the study intervention with the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PF-07940369 and Placebo (Cohort 1) (Experimental): Single dose administration of PF-07940369 and placebo; Within a cohort, participants will receive up to 4 oral doses of PF-07940369 and up to 2 doses of placebo.
  Interventions: Drug: PF-07940369; Drug: Placebo
- PF-07940369 and Placebo (Cohort 2) (Placebo Comparator): Single dose administration of PF-07940369 and placebo; Within a cohort, participants will receive up to 4 oral doses of PF-07940369 and up to 2 doses of placebo.
  Interventions: Drug: PF-07940369; Drug: Placebo

INTERVENTIONS:
Drug: PF-07940369 — Bulk powder for extemporaneous preparation for oral solutions.
Drug: Placebo — Bulk powder for extemporaneous preparation for oral solutions

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and Pharmacokinetics (Pharmacokinetics [PK] to better understand how the drug is changed and eliminated from your body after you take it) of single ascending oral doses of PF-07940369 in healthy adult participants.

This study is seeking participants who:

* are male or female that are not of childbearing potential of 18 years of age or older
* are examined to be healthy

All participants will receive up to 4 single doses of PF-07940369 and up to 2 placebo doses. All treatments will be taken by mouth.

All participants will remain in the study clinic for 4 days for each treatment, for safety review, laboratory collections, and to collect samples for PK.

All participants selected in the study will be required to go through a screening period up to 28 days. A screening period is the time during which a few participants are examined to see whether they are fit for the study. During this period, the participant's medical history and past and current medications will be reviewed. A series of tests will also be performed to see if they are good to be selected for the study. If the participant meets all required criteria and are interested in continuing, the participant will be brought into the study clinic to stay overnight for 4 days for each treatment period. On day 4, the participant will be discharged. About 28 to 35 days after discharge following the final treatment, the participant will be contacted for a follow up visit either in person or by telephone. This is to check up on how the participant is doing and to conclude the study.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

-Male participants and female participants who are not of childbearing potential who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, blood pressure, pulse rate and standard 12 lead ECG.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any of the following conditions: History of iron storage diseases such as hemochromatosis. History of iron utilization disorder such as sideroblastic anemia. Diagnosis of hemolytic anemia or hemoglobinopathy (eg thalassemia). Diagnosis of iron deficiency anemia within 3 months prior to screening. Recent blood donation (within 60 days prior to first dose).
* History of intravenous iron therapy, erythropoiesis stimulating agent therapy (eg erythropoietin) and/or oral iron containing concomitant medications or nutritional supplements exceeding recommended dietary allowances for iron in adults (adult men age 19-50 years: 8 mg, adult women 19-50 years: 18 mg, adults >50 years: 8 mg on weekly average in the 4 weeks prior to randomization).
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥ 140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* An eGFR <90 mL/min/1.73m², as determined by the CKD-EPI equation using Screat calculated using the recommended formulas
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate- age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third- degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening and prior to dosing in each period, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: ALT, AST, Bilirubin ≥1.05 x ULN. Participants with an elevated total bilirubin consistent with Gilberts Disease may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN. Hb <LLN. Serum ferritin < lower limit of the reference range or > upper limit of the reference range for the respective gender and (if applicable) menopausal status. High sensitivity CRP ≥ 3x upper limit of the reference range, if suspected by the investigator to be indicative of inflammation. Albuminuria as defined by urine albumin/creatinine ratio > 30 mg/g. Proteinuria as defined by urine protein/creatinine ratio >200 mg/g. Presence of ≥1+ blood on urine dipstick or red blood cells on urine microscopy. A single repeat assessment for urine dipstick is allowed and, if negative, prior dipstick result will not be exclusionary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline (Day 0) up to 35 days after last dose of study medication
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline up to Day 4
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to Day 4
Number of Participants With Clinically Significant Change From Baseline in Telemetry Findings | Baseline up to Day 4
Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Findings | Baseline up to Day 4

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) of PF-07940369 | Hour 0, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 24, 36, 48, and 72 post-dose in each period
Maximum Observed Plasma Concentration (Cmax) of PF-07940369 | Hour 0, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 24, 36, 48, and 72 post-dose in each period
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07940369 | Hour 0, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 24, 36, 48, and 72 post-dose in each period
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-07940369 | Hour 0, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 24, 36, 48, and 72 post-dose in each period
Plasma Half-Life (t1/2) of PF-07940369 | Hour 0, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 24, 36, 48, and 72 post-dose in each period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5381001